CLINICAL TRIAL: NCT05252702
Title: Aveir Dual-Chamber Leadless i2i IDE Study
Brief Title: Aveir DR i2i Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10416
Record Dates: First submitted 2022-02-09; First posted 2022-02-23 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Pacemaker, Artificial; Cardiac Rhythm Disorder; Bradycardia
Keywords: Bradycardia; Sick Sinus Syndrome; Pacemaker; AV Block; Vasovagal Syncope
MeSH Terms: conditions — Arrhythmias, Cardiac; Bradycardia; Sick Sinus Syndrome; Atrioventricular Block; Syncope, Vasovagal

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, international, single-arm, pivotal investigational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single Arm (Other): Non randomized arm
  Interventions: Device: Aveir DR Leadless Pacemaker System

INTERVENTIONS:
Device: Aveir DR Leadless Pacemaker System — Patients will undergo a dual chamber leadless pacemaker system implant wherein a leadless pacemaker will be implanted in the right ventricle and right atrium

SUMMARY:
Prospective, non-randomized, multi-center, international study designed to evaluate the safety and effectiveness of the Aveir™ Dual-Chamber (DR) Leadless Pacemaker system.

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to evaluate the clinical safety and effectiveness of the Aveir DR Leadless Pacemaker system in a patient population indicated for a DDD(R) pacemaker.

Subjects participating in the study are followed through at least 12 months with data collected at baseline, implant procedure, pre (hospital) discharge, and follow-up at 1 month, 3 months, 6 months, 12 months, and every 6 months thereafter until study completion

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have at least one of the clinical indications before device implant in adherence with ACC/AHA/HRS/ESC dual chamber pacing guidelines
2. Subject is ≥ 18 years of age or age of legal consent, whichever age is greater
3. Subject has a life expectancy of at least one year
4. Subject is willing to comply with clinical investigation procedures and agrees to return to clinic for all required follow-up visits, tests, and exams
5. Subject has been informed of the nature of the clinical investigation, agrees to its provisions and has provided a signed written informed consent, approved by the IRB/EC

Exclusion Criteria:

1. Subject is currently participating in another clinical investigation that may confound the results of this study as determined by the Sponsor
2. Subject is pregnant or nursing and those who plan pregnancy during the clinical investigation follow-up period
3. Subject has presence of anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could confound the assessment of the investigational device and/or implant procedure, limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements of the clinical investigation results
4. Subject has a known allergy or hypersensitivity to < 1 mg of dexamethasone sodium phosphate or any blood or tissue contacting material listed in the IFU
5. Subject has an implanted vena cava filter or mechanical tricuspid valve prosthesis
6. Subject has pre-existing, permanent endocardial pacing or defibrillation leads (does not include lead fragments)
7. Subject has current implantation of either conventional or subcutaneous implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy (CRT) device
8. Subject has an implanted leadless cardiac pacemaker (except for an Aveir ventricular leadless pacemaker)
9. Subject is implanted with an electrically-active implantable medical device with stimulation capabilities (such as neurological or cardiac stimulators)
10. Subject is unable to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 464 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2025-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Harbert, Study Director — Abbott
Locations (78):
- United States (54):
  - HonorHealth, Scottsdale, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - USC University Hospital, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Premier Cardiology, Inc, Newport Beach, California
  - Providence Medical Foundation, Orange, California
  - Huntington Memorial Hospital, Pasadena, California
  - University of California at San Diego (UCSD) Medical Center, San Diego, California
  - Pacific Heart Institute, Santa Monica, California
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Baptist Medical Center, Jacksonville, Florida
  - Naples Heart Rhythm Specialists, PA, Naples, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Prairie Education & Research Cooperative, Springfield, Illinois
  - Iowa Heart Center, West Des Moines, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - Charlton Memorial Hospital, Fall River, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Providence Hospital, Southfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Bryan Heart, Lincoln, Nebraska
  - Catholic Medical Center, Manchester, New Hampshire
  - Jersey Shore University Medical Center, Ocean City, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - New York University Hospital, New York, New York
  - New York Presbyterian Hospital/Cornell University, New York, New York
  - Mount Sinai Hospital, New York, New York
  - New York-Presbyterian/Columbia University Medical Center, New York, New York
  - Cardiac Arrhythmia & Pacemaker Center, Roslyn, New York
  - Wake Forest University Medical Center Clinical Sciences, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital South, Oklahoma City, Oklahoma
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Donald Guthrie Foundation for Education & Research, Sayre, Pennsylvania
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Vanderbilt Heart & Vascular Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia, Austin, Texas
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - Memorial Hermann Hospital, The Woodlands, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Franciscan Heart & Vascular Associates, Tacoma, Washington
  - Aurora Medical Group, Milwaukee, Wisconsin
  - Aspirus Wausau Hospital, Wausau, Wisconsin
- Kepler Universitätsklinikum GmbH, Linz, Upper Austria, Austria
- UZ Gasthuisberg, Leuven, Flemish Brabant, Belgium
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - HSC, Eastern Health, St. John's, Newfoundland and Labrador
  - QE II Health Sciences, Halifax, Nova Scotia
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
- Nemocnice Na Homolce, Prague, Czechia
- France (2):
  - Hopital d'adulte de la Timone, Marseille, Alpes
  - CHRU Albert Michallon, Grenoble
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong, HK SAR
  - Queen Mary Hospital, Hong Kong
- Italy (2):
  - Centro Cardiologico Monzino, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
- Japan (4):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Kurashiki Central Hospital, Kurashiki-shi, Okayama-ken
  - National Cerebral & Cardiovascular Center Hospital, Suita, Osaka
  - Tokyo Women's Medical University, Tokyo
- Amsterdam Academic Medical Centre (AMC), Amsterdam, Netherlands
- Spain (2):
  - Hospital Universitario de Badajoz, Badajoz, Extmdra
  - Hospital Clínic de Barcelona, Barcelona
- National Taiwan University Hospital, Taipei, Taiwan
- United Kingdom (2):
  - John Radcliffe Hospital, Oxford, Soeast
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Any de-identified individual participant data collected will be shared with investigators or other study committee members whose proposed use of the data has been approved by the Aveir DR i2i Study Steering Committee.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available following publication of primary results for 25 years following study completion date.
Access Criteria: Proposals for requesting individual data may be submitted to the Sponsor at AveirDR_IDE@abbott.com.

REFERENCES:
- [Derived] Defaye P, Reddy VY, Ip JE, Doshi RN, Exner DV, Canby RC, Bongiorni MG, Shoda M, Hindricks G, Rashtian MY, Neuzil P, Nevo JR, Badie N, Walker L, Knops RE. Atrioventricular Synchrony Maintained by a Dual-Chamber Leadless Pacemaker in Real-World Conditions. Europace. 2026 Jan 19:euag012. doi: 10.1093/europace/euag012. Online ahead of print. PMID 41554110
- [Derived] Knops RE, Ip JE, Doshi R, Exner DV, Defaye P, Canby R, Bongiorni MG, Shoda M, Hindricks G, Neuzil P, Rashtian M, Breeman KTN, Nevo JR, Ganz L, Hubbard C, Bulusu A, Reddy VY. One-Year Safety and Performance of a Dual-Chamber Leadless Pacemaker. Circ Arrhythm Electrophysiol. 2025 Apr;18(4):e013619. doi: 10.1161/CIRCEP.124.013619. Epub 2025 Mar 27. PMID 40143804
- [Derived] Doshi RN, Ip JE, Defaye P, Reddy VY, Exner DV, Canby R, Shoda M, Bongiorni MG, Hindricks G, Neuzil P, Callahan T, Sundaram S, Booth DF, Richer LP, Badie N, Knops RE. Dual-chamber leadless pacemaker implant procedural outcomes: Insights from the AVEIR DR i2i study. Heart Rhythm. 2025 Sep;22(9):2391-2400. doi: 10.1016/j.hrthm.2025.03.1941. Epub 2025 Mar 13. PMID 40089049
- [Derived] Rashtian MY, Ip JE, Exner DV, Reddy VY, Doshi RN, Defaye P, Canby RC, Bongiorni MG, Shoda M, Hindricks G, Nevo JR, Ligon D, Bulusu A, Knops RE. Temperature-based rate response in a leadless pacemaker system. Heart Rhythm. 2025 Jun;22(6):1533-1540. doi: 10.1016/j.hrthm.2024.11.032. Epub 2024 Nov 22. PMID 39581426
- [Derived] Doshi RN, Ip JE, Defaye P, Exner DV, Reddy VY, Hindricks G, Canby R, Shoda M, Bongiorni MG, Neuzil P, Callahan T, Badie N, Ligon D, Knops RE. Chronic wireless communication between dual-chamber leadless pacemaker devices. Heart Rhythm. 2025 Apr;22(4):1010-1020. doi: 10.1016/j.hrthm.2024.10.020. Epub 2024 Oct 19. PMID 39427688
- [Derived] Knops RE, Reddy VY, Ip JE, Doshi R, Exner DV, Defaye P, Canby R, Bongiorni MG, Shoda M, Hindricks G, Neuzil P, Rashtian M, Breeman KTN, Nevo JR, Ganz L, Hubbard C, Cantillon DJ; Aveir DR i2i Study Investigators. A Dual-Chamber Leadless Pacemaker. N Engl J Med. 2023 Jun 22;388(25):2360-2370. doi: 10.1056/NEJMoa2300080. Epub 2023 May 20. PMID 37212442
- [Derived] Reddy VY, Exner DV, Doshi R, Tomassoni G, Bunch TJ, Friedman P, Estes NAM, Neuzil P, de la Concha JF, Cantillon DJ; LEADLESS II Investigators. 1-Year Outcomes of a Leadless Ventricular Pacemaker: The LEADLESS II (Phase 2) Trial. JACC Clin Electrophysiol. 2023 Jul;9(7 Pt 2):1187-1189. doi: 10.1016/j.jacep.2023.01.031. Epub 2023 Mar 22. No abstract available. PMID 36951813

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject enrollment in the Aveir DR i2i IDE study began on February 2, 2022 in Czech Republic, February 24, 2022 in the US, April 7, 2022 in Canada, October 14, 2022 in Hong Kong, and February 9, 2023 in Taiwan. The study enrolled 464 de novo subjects at 77 sites worldwide
Groups:
- Enrolled de Novo Cohort: The enrolled de novo cohort consisted of subjects that were screened for and met eligibility criteria, provided written informed consent, and were scheduled to undergo a dual chamber Aveir DR leadless pacemaker system implant wherein a leadless pacemaker was to be implanted in the right ventricle and right atrium
Period: Overall Study
Arm/Group | Enrolled de Novo Cohort
Started (Enrolled subjects) | 464
Attempted Implant | 452
Predischarge Visit | 450
1-month Visit | 443
3-month Visit | 442
6-month Visit | 435
12-month Visit | 360
18-month Visit | 100
Completed (24-month Visit) | 30
Not Completed | 434
Not completed — No attempted implant, subjects withdrawn | 12
Not completed — Death | 16
Not completed — System explant | 5
Not completed — Lost to Follow-up | 1
Not completed — Withdrawn by investigator | 1
Not completed — Visit not due | 306
Not completed — Visit within window but not completed | 92
Not completed — Unsuccessful implant | 1

BASELINE CHARACTERISTICS:
Groups:
- Enrolled de Novo Cohort With Attempted Implant: The enrolled de novo cohort with attempted implant group consisted of subjects that were screened for and met eligibility criteria, provided written informed consent, and had an attempted dual chamber Aveir DR leadless pacemaker system implant
Arm/Group | Enrolled de Novo Cohort With Attempted Implant
Number analyzed (Participants) | 452
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174
  Male | 278
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1
  Asian | 46
  Black or African American | 13
  White | 282
  Declined/Unable to Disclose | 104
  Unknown | 5
  Multi-Racial | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 331
  Declined/Unable to Disclose | 100
  Unknown | 6
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 11
  United States | 280
  Czechia | 33
  Japan | 24
  United Kingdom | 8
  Spain | 18
  Canada | 33
  Austria | 5
  Netherlands | 4
  Belgium | 6
  Taiwan | 5
  Italy | 7
  France | 18
Height [Mean (Standard Deviation); unit: cm] | 170.7 (10.8)
Weight [Mean (Standard Deviation); unit: kg] | 81.6 (19.8)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Free From Aveir DR System-Related Complications at 3-months
Description: Aveir DR Leadless Pacemaker system complication-free-rate in de novo subjects. A complication was defined as a device-or-procedure-related serious adverse event. Complications included Atrial LP, Ventricular LP, and implant procedure-related complications. Complications possibly related or related to COVID-19 were excluded.
Time Frame: 3 months
Population: The primary analysis population for the primary safety endpoint was based on subjects in the full analysis population. The full analysis population included the first 300 consecutive de novo subjects who provided written informed consent and had an attempted implant. A de novo subject was a subject who did not have an implanted pacemaker on the date of consent through the date of the attempted Aveir LP implant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Primary Analysis Population: The first 300 consecutive de novo subjects who provided written informed consent and had an attempted implant.
Arm/Group | Primary Analysis Population
Number analyzed (Participants) | 300
percentage of participants | 90.3 [87 to 93.7]
Statistical Analysis 1: Comparison: Primary Analysis Population; Test type: Superiority — The primary safety endpoint hypothesis at 3 months was formally expressed as: H0: CFR ≤ 78% vs. H1: CFR > 78% where 78% was the performance goal (PG); p < 0.0001, one-sided Z-test — The CFR was estimated as a binomial proportion and a one-sided 97.5% lower confidence bound of the CFR was calculated using the normal approximation. The null hypothesis was to be rejected at the 2.5% significance level if the LCB exceeded the PG; The p-value from a one-sided Z-test for the binomial proportion was calculated and compared to the 0.025 significance level; binomial proportion = 90.3, 97.5% CI 1-sided [lower limit 87]

2. Primary Outcome: Percentage of Participants Free From Aveir DR System-Related Complications at 12-months
Description: as for outcome 1
Time Frame: 12 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Analysis Population
Number analyzed (Participants) | 300
percentage of participants | 88.6 [84.5 to 91.8]
Statistical Analysis 1: Comparison: Primary Analysis Population; Test type: Superiority — The primary safety endpoint hypothesis at 12 months was formally expressed as: H0: CFR ≤ 76.5% vs. H1: CFR > 76.5% where 76.5% is the performance goal. The CFR was estimated using a Kaplan-Meier survival analysis and the 97.5% lower confidence bound of CFR was calculated using the Greenwood variance estimates; p < 0.0001, one-sided Z-test — The null hypothesis was to be rejected at the 2.5% significance level if the LCB exceeded the Performance Goal (PG) of 76.5%; The p-value for the one-sided Z-test was calculated and compared to the 2.5% significance level; Kaplan-Meier = 88.6, 97.5% CI 1-sided [lower limit 84.5]

3. Primary Outcome: Percentage of Subjects With Acceptable Atrial Threshold and Amplitude Measurements at 3-months
Description: Composite success rate of acceptable atrial pacing thresholds and P-wave amplitudes in de novo subjects. A subject was considered to have met the primary effectiveness endpoint #1 if the pacing threshold voltage was ≤ 3.0 V at 0.4 ms at the 3-month visit and the sensed P-wave amplitude was ≥ 1.0 mV at the 3-month visit.
Time Frame: 3 months
Population: Among the 300 subjects in the full analysis population, 3 subjects were excluded due to unsuccessful atrial device implant and unmeasurable p-wave amplitude.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Analysis Population
Number analyzed (Participants) | 297
percentage of participants | 90.8 [87.5 to 94.1]
Statistical Analysis 1: Comparison: Primary Analysis Population; The primary effectiveness endpoint #1 hypothesis at 3 month was formally expressed as: H0: Rate ≤ 82.5% vs. H1: Rate > 82.5% where 82.5% was the performance goal (PG); Test type: Superiority; p < 0.0001, one-sided Z-test — The null hypothesis was to be rejected at the 2.5% significance level if the LCB exceeded the PG of 82.5%; The p-value for the one-sided Z-test was to be calculated and compared to the 2.5% significance level; binomial proportion = 90.8, 97.5% CI 1-sided [lower limit 87.5]

4. Primary Outcome: Percentage of Subjects With Acceptable Atrial Threshold and Amplitude Measurements at 12-months
Description: Composite success rate of acceptable atrial pacing thresholds and P-wave amplitudes in de novo subjects. A subject was considered to have met the success criteria for the endpoint if the pacing threshold voltage was ≤ 3.0 V at 0.4 ms at the 12-month visit and the sensed P-wave amplitude was ≥ 1.0 mV at the 12-month visit.
Time Frame: 12 months
Population: Out of 300 subjects, 8 subjects were excluded from primary effectiveness endpoint. 2 were excluded for unsuccessful atrial device implant and 6 were excluded due to unmeasurable P-wave amplitudes and pacing voltages at the 12-month visit due to atrial fibrillation/ atrial tachycardia.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Analysis Population
Number analyzed (Participants) | 292
percentage of participants | 92.8 [89.7 to 95.8]
Statistical Analysis 1: Comparison: Primary Analysis Population; The primary effectiveness endpoint #1 hypothesis at 12 months was formally expressed as: H0: Rate ≤ 80% vs. H1: Rate > 80% where 80% was the performance goal (PG); Test type: Superiority; p < 0.0001, one-sided Z-test — The null hypothesis was to be rejected at the 2.5% significance level if the LCB exceeded the PG of 80%; The p-value for the one-sided Z-test was to be calculated and compared to the 2.5% significance level; binomial proportion = 92.8, 97.5% CI 1-sided [lower limit 89.7] — The Rate at 12 months was estimated as a binomial proportion and the one-sided 97.5% LCB of the Rate was calculated using the normal approximation

5. Primary Outcome: Percentage of Participants With AV Synchrony Success Rate at Rest While Seated
Description: AV synchrony success was defined as subjects with a paced or sensed ventricular beat within 300 ms following a paced or sensed atrial beat (i.e., a synchronous cycle) for at least 70% of evaluable cardiac cycles.
Time Frame: 3 months
Population: Out of 300 subjects in the full analysis population, 2 were excluded due to unsuccessful atrial implants. Then out of 298 subjects, 277 subjects with AV Synchrony data available to define endpoint success were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Analysis Population
Number analyzed (Participants) | 277
percentage of participants | 98.2 [96.6 to 99.8]
Statistical Analysis 1: Comparison: Primary Analysis Population; The primary effectiveness endpoint #2 hypothesis was formally expressed as: H0: RateAV ≤ 83% vs. H1: RateAV > 83% where 83% is the performance goal; Test type: Superiority; p < 0.0001, one-sided Z-test — The null hypothesis was to be rejected at the 2.5% significance level if the LCB exceeded the PG of 83%; The p-value for the one-sided Z-test was to be calculated and compared to the 2.5% significance level; binomial proportion = 98.2, 97.5% CI 1-sided [lower limit 96.6]

6. Secondary Outcome: Percentage of Participants Free From Aveir Atrial Leadless Pacemaker-Related Complications at 3-months
Description: The secondary safety endpoint evaluated a 3-month Atrial LP related complication-free rate based on CEC adjudication of adverse events. An Atrial LP complication was defined as an atrial device-or-procedure-related serious adverse event. Complications that were exclusively related to the Ventricular LP or its delivery/retrieval were not considered Atrial LP complications and were excluded from the evaluation. For a conservative approach, complications that could not exclusively be determined to be related to the ventricular or Atrial LP were still considered Atrial LP complications. For example, procedure-related femoral access complications were adjudicated as Atrial LP complications.
Time Frame: 3 months
Population: The primary analysis population for the secondary safety endpoint was based on subjects in the full analysis population, which included the first 300 consecutive de novo subjects who provided written informed consent and had an attempted implant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Analysis Population
Number analyzed (Participants) | 300
percentage of participants | 91.3 [88.1 to 94.5]
Statistical Analysis 1: Comparison: Primary Analysis Population; The secondary safety endpoint hypothesis at 3 months was formally expressed as: H0: CFRA ≤ 84% vs. H1: CFRA > 84% where 84% was the performance goal; Test type: Superiority; p = 0.0003, one-sided Z-test — The null hypothesis was to be rejected at the 2.5% significance level if the lower confidence bound exceeded the Performance Goal (PG) of 84%; The p-value from a one-sided Z-test for the binomial proportion was to be calculated and compared to the 0.025 significance level; binomial proportion = 91.3, 97.5% CI 1-sided [lower limit 88.1]

7. Secondary Outcome: Percentage of Participants Free From Aveir Atrial Leadless Pacemaker-Related Complications at 12-months
Description: The secondary safety endpoint analysis evaluated the 12-month Atrial LP related complication-free rate (CFRA) based on CEC adjudication of adverse events. An Atrial LP complication was defined as an atrial device-or-procedure-related serious adverse event. Complications that were exclusively related to the Ventricular LP or its delivery/retrieval were not considered Atrial LP complications and were excluded from the evaluation. For a conservative approach, complications that could not exclusively be determined to be related to the ventricular or Atrial LP were still considered Atrial LP complications. For example, procedure-related femoral access complications were adjudicated as Atrial LP complications. Complications possibly related or related to COVID-19 were excluded.
Time Frame: 12 months
Population: The analysis population for the secondary safety endpoint was based on subjects in the full analysis population, which included the first 300 consecutive de novo subjects who provided written informed consent and had an attempted implant.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Analysis Population
Number analyzed (Participants) | 300
percentage of participants | 91.0 [87.1 to 93.7]
Statistical Analysis 1: Comparison: Primary Analysis Population; The secondary safety endpoint hypothesis at 12 months was formally expressed as: H0: CFRA ≤ 82% vs. H1: CFRA > 82% where 82% is the performance goal; Test type: Superiority; p < 0.0001, one-sided Z-test — The null hypothesis was to be rejected at the 2.5% significance level if the LCB exceeded the Performance Goal (PG) of 82%; The p-value for the one-sided Z-test was to be calculated and compared to the 2.5% significance level; Kaplan-Meier = 91.0, 97.5% CI 1-sided [lower limit 87.1], Standard Error of Mean 1.7 — The 97.5% lower confidence bound (LCB) of CFRA was calculated using the Greenwood variance estimates

8. Secondary Outcome: Slope of the Normalized Increase in the Sensor Indicated Rate Versus Normalized Workload of the Aveir Atrial Leadless Pacemaker During Exercise Testing
Description: Appropriate and proportional rate response of the Aveir Atrial Leadless Pacemaker in de novo subjects was tested during staged exercise testing. Exercise test data provided an estimate of the slope of the normalized increase in sensor-indicated rate versus normalized workload for each subject. Normalizing a variable eliminates the unit and expresses it from 0-1.0. Since both axes are normalized sensor rate and workload, there is no distinct unit of measure. Values on the vertical axis are derived from the difference of the sensor indicated rate at each exercise stage and the base rate, divided by the difference of the age-predicted maximum heart rate and base rate. Values on the horizontal axis are derived from the difference in the workload at each exercise stage and resting workload, divided by the difference of the maximum achieved workload and resting workload. A slope value of 1.0 indicates the pacemaker's sensor-indicated rate increases linearly with an increase in workload.
Time Frame: 3 months
Population: Subjects with Analyzable CAEP Data
Measure: Mean (95% Confidence Interval); unit: unitless
Groups:
- Chronotropic Assessment Exercise Protocol (CAEP) Group: Data from subjects who had completed the 6MWT protocol and had completed at least stage 3 of the CAEP exercise protocol, or 3.6 metabolic equivalent of task (METs), were included in the analysis.
Arm/Group | Chronotropic Assessment Exercise Protocol (CAEP) Group
Number analyzed (Participants) | 20
unitless | 0.91 [0.78 to 1.04]
Statistical Analysis 1: Comparison: Chronotropic Assessment Exercise Protocol (CAEP) Group; An analysis of these data provided an estimate of the 95% confidence interval for the mean slope across analyzable subjects, which had a pre-specified success criterion requiring that this confidence interval must fall between slopes of 65% and 135%. The following hypothesis was evaluated: H0: Mean Slope < 0.65 or Mean Slope > 1.35 H1: 0.65 ≤ Mean Slope ≤ 1.35; Test type: Other; p < 0.001, t-test, 1 sided; Two one-sided t-tests (TOST), with an alpha level of 0.025, and n-1 degrees of freedom; mixed effects model for repeated measure = 0.91, 95% CI 2-sided [0.78 to 1.04], Standard Error of Mean 0.06

ADVERSE EVENTS:
Time Frame: From implant attempt to last subject follow-up, ranging from 0 to 24 months
Description: Adverse event data includes both device and non-device related events.
Arm/Group | Enrolled de Novo Cohort With Attempted Implant
All-Cause Mortality (participants affected / at risk) | 16/452
Serious Adverse Events (participants affected / at risk) | 202/452
Other Adverse Events (participants affected / at risk) | 366/452
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled de Novo Cohort With Attempted Implant (N=452)
Cardiac Arrhythmia - Atrial Fibrillation (Cardiac disorders) | 41 (44)
Heart Failure (Cardiac disorders) | 18 (22)
Cardiac Arrhythmia - Supraventricular Arrhythmia (Cardiac disorders) | 11 (14)
Infection, Local at Access Site, or Systemic (Infections and infestations) | 10 (12)
Syncope (General disorders) | 3 (7)
Accidental Injury/Mechanical Trauma (Injury, poisoning and procedural complications) | 6 (6)
Pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Respiratory Failure/Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Electrolyte Disbalance (Investigations) | 3 (5)
Urinary Tract Infection/UTI (Renal and urinary disorders) | 4 (5)
Chest Pain - Non-Cardiac (General disorders) | 5 (5)
Death (General disorders) | 5 (5)
Sepsis (Infections and infestations) | 5 (5)
Stroke (Nervous system disorders) | 5 (5)
Covid-19 Infection (Infections and infestations) | 5 (5)
Hypotension (Cardiac disorders) | 4 (4)
Malignant Tumor/Malignant Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Myocardial Infarction (Cardiac disorders) | 4 (4)
Renal Failure/Insufficiency (Renal and urinary disorders) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 2 (3)
Peripheral Artery Disease (Vascular disorders) | 2 (3)
Dyspnea (General disorders) | 3 (3)
Transient Ischemic Attack (Cardiac disorders) | 3 (3)
Valve Disease (Cardiac disorders) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Angina Pectoris (Cardiac disorders) | 2 (2)
Cardiac Perforation (Cardiac disorders) | 3 (3)
Coronary Artery Disease (Cardiac disorders) | 2 (2)
Diabetes (Endocrine disorders) | 2 (2)
Gastrointestinal Bleeding/Hemorrhage (Gastrointestinal disorders) | 2 (2)
Hernia (Musculoskeletal and connective tissue disorders) | 2 (2)
Hypertension (Cardiac disorders) | 2 (2)
Hypoglycemia (Blood and lymphatic system disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2)
Pre-Syncope (General disorders) | 3 (3)
Thrombosis (Injury, poisoning and procedural complications) | 3 (3)
Weakness (General disorders) | 2 (2)
Cardiac Arrhythmia - Ventricular Arrhythmia (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Dizziness (General disorders) | 6 (6)
Encephalopathy (Nervous system disorders) | 1 (1)
Excessive Bleeding (Injury, poisoning and procedural complications) | 1 (1)
Gallbladder Disease (Hepatobiliary disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Hematoma Formation, Including Retroperitoneal Hematoma/Hemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Pneumothorax/Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Reaction/Toxic Effect Due to Contrast Media (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 6 (6)
Cholecystitis (Hepatobiliary disorders) | 4 (4)
Altered Mental Status (Psychiatric disorders) | 3 (3)
Cardiac Arrest (Cardiac disorders) | 3 (3)
Femur Fracture (Injury, poisoning and procedural complications) | 3 (3)
Fluid Overload (Injury, poisoning and procedural complications) | 3 (3)
Parkinson's Disease (Nervous system disorders) | 3 (3)
Mechanical Device Dislodgement (Injury, poisoning and procedural complications) | 3 (3)
Pulmonary Hypertension (Cardiac disorders) | 2 (2)
Shock (Infections and infestations) | 2 (2)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1)
Acute Hepatitis (Infections and infestations) | 1 (1)
Acute Psychosis (Psychiatric disorders) | 1 (1)
Adjustment Disorder (Psychiatric disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Anal Nodule (General disorders) | 1 (1)
Av Fistula Malfunction (Blood and lymphatic system disorders) | 1 (1)
Calciphylaxis of Penis Fistula (Blood and lymphatic system disorders) | 1 (1)
Carotid Artery Stenosis (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Cerebrovascular Accident (Vascular disorders) | 1 (1)
Chest Pain Unspecified (General disorders) | 1 (1)
Chronic Right Elbow Olecranon Bursitis (General disorders) | 1 (1)
Coxarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cystitis (Hepatobiliary disorders) | 1 (1)
Diarrhea (Hepatobiliary disorders) | 1 (1)
Enlarged Prostate (Reproductive system and breast disorders) | 1 (1)
Gastroesophageal Reflux (Gastrointestinal disorders) | 1 (1)
Generalized Weakness (General disorders) | 1 (1)
Gonarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Head Laceration (Injury, poisoning and procedural complications) | 1 (1)
Hyponatremia (Investigations) | 1 (1)
Ileitis (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Knee Arthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Left Atrial Appendage Occlusion (Blood and lymphatic system disorders) | 1 (1)
Leg Weakness (General disorders) | 1 (1)
Low Ejection Fraction (Cardiac disorders) | 1 (1)
Lumbar Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Parotid Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pseudophakia (Eye disorders) | 1 (1)
Sacroiliac Join Dysfunction (Musculoskeletal and connective tissue disorders) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Stent Restenosis (Cardiac disorders) | 1 (1)
Suicidal Ideations (Psychiatric disorders) | 1 (1)
Thyroid Nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Vertebrae Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Vertigo (General disorders) | 1 (1)
Vision Loss (Eye disorders) | 1 (1)
Vomiting (General disorders) | 1 (1)
Threshold Elevation (General disorders) | 7 (7)
Inadequate Fixation During Implant with LP Migration (Injury, poisoning and procedural complications) | 5 (5)
Urinary Retention (Renal and urinary disorders) | 5 (5)
Inadequate Fixation During Implant Without LP Migration (Injury, poisoning and procedural complications) | 3 (4)
Pericardial Effusion or Rub (Cardiac disorders) | 4 (4)
Access Site Bleeding (Injury, poisoning and procedural complications) | 3 (3)
Intermittent Capture (Injury, poisoning and procedural complications) | 2 (2)
Tricuspid Valve Damage And/or Regurgitation (Cardiac disorders) | 1 (1)
Pacemaker Syndrome (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 9 (10)
Intermittent or Loss of I2i Communication (Injury, poisoning and procedural complications) | 1 (1)
Oversensing (Injury, poisoning and procedural complications) | 3 (3)
Arteriovenous Fistula (Vascular disorders) | 1 (1)
Pleural Effusion (Blood and lymphatic system disorders) | 1 (1)
Pulmonary Embolism (Blood and lymphatic system disorders) | 1 (1)
Cardiac Tamponade (Cardiac disorders) | 1 (1)
Inability to Release and Redock the LP (Injury, poisoning and procedural complications) | 1 (1)
False Magnet Mode (Injury, poisoning and procedural complications) | 1 (1)
Cardiopulmonary Arrest (Cardiac disorders) | 1 (1)
Access site Oozing (Injury, poisoning and procedural complications) | 1 (1)
Arterial Laceration (Injury, poisoning and procedural complications) | 1 (1)
Cardiogenic Shock (Infections and infestations) | 1 (1)
Complete Heart Block (Cardiac disorders) | 1 (1)
Device Dislogdement (Injury, poisoning and procedural complications) | 12 (14)
Complete AV Block (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled de Novo Cohort With Attempted Implant (N=452)
Pain (Musculoskeletal and connective tissue disorders) | 34 (41)
Cardiac Arrhythmia - Atrial Fibrillation (Cardiac disorders) | 37 (40)
Palpitations (Cardiac disorders) | 34 (36)
Covid-19 Infections (Infections and infestations) | 27 (27)
Dizziness (General disorders) | 29 (30)
Infection, Local at Access Site, or Systemic (Infections and infestations) | 21 (25)
Urinary Tract Infection/UTI (Renal and urinary disorders) | 13 (16)
Chest Pain - Non-Cardiac (General disorders) | 17 (19)
Dyspnea (General disorders) | 25 (25)
Accidental Injury/Mechanical Trauma (Injury, poisoning and procedural complications) | 12 (14)
Hypotension (Cardiac disorders) | 11 (13)
Heart Failure (Cardiac disorders) | 12 (15)
Cardiac Arrhythmia - Supraventricular Arrhythmia (Cardiac disorders) | 12 (13)
Syncope (General disorders) | 7 (8)
Hypertension (Cardiac disorders) | 8 (8)
Abdominal Pain (General disorders) | 6 (7)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Renal Failure/Insufficiency (Renal and urinary disorders) | 7 (7)
Angina Pectoris (Cardiac disorders) | 5 (5)
Cardiac Arrhythmia - Ventricular Arrhythmia (Cardiac disorders) | 6 (6)
Electrolyte Disbalance (Investigations) | 5 (5)
Weakness (General disorders) | 8 (8)
Constipation (Gastrointestinal disorders) | 3 (3)
Nausea (General disorders) | 3 (3)
Pleural Effusion (Blood and lymphatic system disorders) | 3 (3)
Dehydration (Investigations) | 2 (2)
Hernia (Musculoskeletal and connective tissue disorders) | 2 (2)
Pulmonary Edema (Cardiac disorders) | 4 (4)
Urinary Retention (Renal and urinary disorders) | 3 (3)
Valve Disease (Cardiac disorders) | 2 (2)
Access Site Bleeding Event (Injury, poisoning and procedural complications) | 23 (23)
Aortic Aneurysm (Cardiac disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Coronary Artery Disease (Cardiac disorders) | 1 (1)
Diabetes (Endocrine disorders) | 1 (1)
Gastrointestinal Bleeding/Hemorrhage (Gastrointestinal disorders) | 1 (1)
Groin Pain (Reproductive system and breast disorders) | 2 (2)
Hypoglycemia (Blood and lymphatic system disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Oversensing (Injury, poisoning and procedural complications) | 1 (1)
Pericardial Effusion or Rub (Cardiac disorders) | 5 (5)
Peripheral Artery Disease (Blood and lymphatic system disorders) | 1 (1)
Pre-Syncope (General disorders) | 1 (1)
Thrombosis (Injury, poisoning and procedural complications) | 2 (2)
Transient Ischemic Attack (Cardiac disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 10 (10)
Anxiety (Psychiatric disorders) | 3 (5)
Diarrhea (General disorders) | 5 (5)
Headache (General disorders) | 4 (4)
Hematuria (Renal and urinary disorders) | 4 (4)
Lower Extremity Edema (Blood and lymphatic system disorders) | 5 (5)
Fatigue (General disorders) | 5 (5)
Acute Kidney Injury (Renal and urinary disorders) | 4 (4)
Asthenia (General disorders) | 3 (3)
Depression (Psychiatric disorders) | 3 (3)
Pre-Syncope (General disorders) | 2 (2)
Shortness of Breath (General disorders) | 2 (2)
Chest Pain - Unspecified (Musculoskeletal and connective tissue disorders) | 4 (4)
Cough (General disorders) | 2 (2)
Dementia (Nervous system disorders) | 2 (2)
Elevated D-Dimer (Blood and lymphatic system disorders) | 2 (2)
Fever (Infections and infestations) | 2 (2)
Infection (Infections and infestations) | 2 (2)
Skin Lesions (Skin and subcutaneous tissue disorders) | 2 (2)
Skin Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Thyroid Leves Abnormal (Endocrine disorders) | 2 (2)
Adjustment Disorder (Psychiatric disorders) | 1 (1)
Allergic Reaction (General disorders) | 2 (2)
Altered Mental State (Psychiatric disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Asteatosis Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Asthmatic Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Barrett's Esophagus (Gastrointestinal disorders) | 1 (1)
Bilateral Upper Limb Numbness (Musculoskeletal and connective tissue disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Bruise (Injury, poisoning and procedural complications) | 1 (1)
Cardiomegaly (Cardiac disorders) | 1 (1)
Carpal Tunnel Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Chest Discomfort (General disorders) | 2 (2)
Chest Pain Unspecified (General disorders) | 1 (1)
Chest Pressure (General disorders) | 1 (1)
Chest TIghtness (General disorders) | 1 (1)
Chronic Dislocated Right Shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Cirrhotic Liver (Hepatobiliary disorders) | 1 (1)
Coccyx Fracture (Injury, poisoning and procedural complications) | 1 (1)
Confusion (General disorders) | 1 (1)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1 (1)
Deterioration of Vision (Eye disorders) | 1 (1)
Drug-Induced Parkinsonism (Nervous system disorders) | 1 (1)
Dysautonomia (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Nervous system disorders) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1)
Exacerbation of Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eye Floaters (Eye disorders) | 1 (1)
Eye Irritation (Eye disorders) | 1 (1)
Fistula Discharge (General disorders) | 1 (1)
Fluid Overload (Blood and lymphatic system disorders) | 1 (1)
Frontoparietal Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastroesophageal Reflux (Gastrointestinal disorders) | 1 (1)
Hallucination (General disorders) | 1 (1)
Heartburn (General disorders) | 1 (1)
Hepatic Lesion (Hepatobiliary disorders) | 1 (1)
Hot Flashes (General disorders) | 1 (1)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyponatremia (Investigations) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Ingrown Toenail (Skin and subcutaneous tissue disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Left Arm Fracture (Injury, poisoning and procedural complications) | 1 (1)
Left Hand Numbness (General disorders) | 1 (1)
Leg Weakness (General disorders) | 1 (1)
Low Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Lung Nodules (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malaise (General disorders) | 1 (1)
Nodules Right Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Numbness/Tingling in Lower (General disorders) | 1 (1)
Ophthalmic Herpes Zoster (Infections and infestations) | 1 (1)
Oral Ulcers (Infections and infestations) | 1 (1)
Orthostatic Hypotension (General disorders) | 1 (1)
Pacemaker Mediated Tachycardia (Cardiac disorders) | 5 (5)
Pain (General disorders) | 1 (1)
Pansinusitis (Infections and infestations) | 1 (1)
Paresthesia (General disorders) | 1 (1)
Patent Foramen Ovale (Cardiac disorders) | 1 (1)
Periodontal Disease (General disorders) | 1 (1)
Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Post-Operative Wound Infection (Infections and infestations) | 1 (1)
Pressure in the Head (General disorders) | 1 (1)
Pressure Ulcer (General disorders) | 1 (1)
Pruritus (General disorders) | 2 (2)
Pulmonary Nodules (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Qt Prolongation (Cardiac disorders) | 1 (1)
Rapid Heart Rate (Cardiac disorders) | 1 (1)
Rectal Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Restless Leg Syndrome (General disorders) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1)
Right Second Toe Blister (Injury, poisoning and procedural complications) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Seizure (General disorders) | 1 (1)
Skin Cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Stasis Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Sublingual Bleeding (Injury, poisoning and procedural complications) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombophlebitis (Blood and lymphatic system disorders) | 1 (1)
Thyroglossal Duct Cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tinea Cruris (Infections and infestations) | 1 (1)
Tongue Laceration (Injury, poisoning and procedural complications) | 1 (1)
Tympan Perforation (Injury, poisoning and procedural complications) | 1 (1)
Ulcerative Colitis (Hepatobiliary disorders) | 1 (1)
Unsteady Gait (Gastrointestinal disorders) | 1 (1)
Urinary Hesitancy (Renal and urinary disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Varicose Veins (Blood and lymphatic system disorders) | 1 (1)
Vein Stenosis (Blood and lymphatic system disorders) | 1 (1)
Venous Disease (Blood and lymphatic system disorders) | 1 (1)
Venous Reflux (Blood and lymphatic system disorders) | 1 (1)
Vision Loss (Eye disorders) | 1 (1)
Vomiting (General disorders) | 1 (1)
Wrist Sprain (Injury, poisoning and procedural complications) | 1 (1)
Threshold Elevation (General disorders) | 22 (23)
Intermitted or Loss of I2i Communication (Injury, poisoning and procedural complications) | 16 (16)
Hematoma Formation, Including Retroperitoneal Hematoma/Hemorrhage (Injury, poisoning and procedural complications) | 14 (14)
Inability to Interrogate or Program due to Programmer or LP Malfunction (Injury, poisoning and procedural complications) | 9 (11)
Phrenic Nerve/Diaphragmatic/Extra-Cardiac Stimulation (Nervous system disorders) | 3 (4)
Intermittent Capture (Injury, poisoning and procedural complications) | 2 (3)
Pacemaker Syndrome (Cardiac disorders) | 3 (3)
Failure to Capture/Loss of Capture (Injury, poisoning and procedural complications) | 2 (2)
Tricuspid Valve Damage and/or Regurgitation (Cardiac disorders) | 2 (2)
Interruption of Desired LP Function due to Electrical Interference, Electromyogenic or Electromagnet (Injury, poisoning and procedural complications) | 1 (1)
Undersensing (Injury, poisoning and procedural complications) | 1 (1)
False Magnet Mode (Injury, poisoning and procedural complications) | 7 (7)
Intermittent or Loss of Sensing (Injury, poisoning and procedural complications) | 1 (1)
Access Site Induration (Injury, poisoning and procedural complications) | 1 (1)
Access Site Oozing (Injury, poisoning and procedural complications) | 1 (1)
Vascular Dissection (Vascular disorders) | 1 (1)
Inability to Release and Redock the LP (Injury, poisoning and procedural complications) | 2 (2)
Non-Healing Wound (Injury, poisoning and procedural complications) | 2 (2)
Inability to Interrogate Device Due to Interference from Swan Ganz Continuous Cardiac Output Monitor (Injury, poisoning and procedural complications) | 1 (1)
Left Ventricular Dysfunction (Cardiac disorders) | 1 (1)
LP Found in Rom Mode (Injury, poisoning and procedural complications) | 1 (1)
Access Site Infection (Infections and infestations) | 1 (1)
Epistaxis (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Radial Artery Occlusion (Vascular disorders) | 1 (1)
Visual Hallucinations (General disorders) | 1 (1)
Right Bundle Branch Block (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Clinical Investigation Plan (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/02/NCT05252702/Prot_000.pdf
  • Study Protocol: Clinical Investigation Plan for Europe (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/02/NCT05252702/Prot_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/02/NCT05252702/SAP_002.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan for Europe (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT05252702/SAP_003.pdf